CLINICAL TRIAL: NCT03827135
Title: Effects of Cyriax Manipulation in Cervical Discogenic Pain
Brief Title: Cyriax Manipulation in Cervical Discogenic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Aisha Razzaq
Record Dates: First submitted 2019-01-27; First posted 2019-02-01 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Cervical Discogenic Pain (Disorder)
Keywords: Cervical Discogenic pain; Cyriax manipulation; Neck Pain Disability index

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): Cervical isometrics and Muscle Stretching
  Interventions: Other: Traditional physical therapy
- Cyriax manipulation (Experimental): Experimental group was given cyriax manipulation protocol along with the cervical isometrics and muscle stretching.
  Interventions: Other: Cyriax manipulation

INTERVENTIONS:
Other: Traditional physical therapy — Cervical isometrics 10 repetitions×1 set, 4 days/week and targeted muscle strechings (trapezius, scalenes and sternocleidomastoid) 10 repetitions×1 set, 4 days/week.
  Total of 4 sessions were given each consisting of 40 mins.
  Arms: Traditional physical therapy
Other: Cyriax manipulation — Experimental group was given cyriax manipulation protocol along with the cervical isometrics and muscle strechings.
  Traction with rotation was not given in cases of bilateral arm pain. cervical isometrics 10 repetitions×1 set, 4 days/week and targeted muscle strechings (trapezius, scalenes and sternocleidomastoid) 10 repetitions×1 set, 4 days/week.
  Total of 4 sessions were given each consisting of 40 mins.
  Arms: Cyriax manipulation

SUMMARY:
The aim of this research is to find and compare the effect of traditional physical therapy and Cyriax manipulation on pain, range of motion and disability in patients with cervical discogenic pain. Randomized controlled trials done at Benazir Bhutto hospital, Rawalpindi . The sample size was 40. The subjects were divided in two groups, 20 subjects in traditional physical therapy group and 20 in Cyriax manipulation group. Study duration was of 6 months. Sampling technique applied was purposive non probability sampling technique. Only 25-45 years individual with cervical discogenic pain were included. Tools used in the study are Numeric pain rating scale (NPRS) and neck disablity index (NDI). Data was be analyzed through SPSS 21.

DETAILED DESCRIPTION:
Cervical disc displacement is a significant cause of neck and arm pain and disability in majority of individuals. It causes a great burden on physical, social and emotional quality of life of patients. The cervical disc herniation is characterized by prolapsed nucleus pulposus material through the annulus into the spinal canal. The local mechanical or chemical irritation of neural structures typically leads to symptoms of radiculopathy, head and neck pain or myelopathy. The disc bulge may be postero-central to compress the dura matter, causing multi segmental pain and affect the scapular area. It can also be postero-lateral causing the root signs, that have dermatomal behavior and affect the upper limb in specific pattern. Postero-central bulge can also shift to postero-lateral with symptoms shifting from centralization to radiculopathy.

The State of U.S. Health: Burden of Diseases, Injuries and Risk Factors describes cervical pain among 5 most contributing factor in causing years lived in disability. the ratio tremendously increases after 40 years. Studies describing impact of chronic neck pain on general health care reveals 14% of patients reports grade II to grade IV neck pain with high pain intensity and disability.

Disc displacement disorders are included among the mechanical causes of neck pain. Symptomatic disc displacements can occur at any age but have different clinical features depending on the age group. In young adults nucleus pulposus can involve which is rare in old age. Diagnoses can be established on clinical findings along with patient's history and the functional examination. Disc displacement can occur in postero-central and Postero- lateral displacement. Movement of the disc posteriorly causes stress on the posterior longitudinal ligament and also on the anterior part of the Dura mater. As a result of this the pain travels in more than one segment with dural reference. Pain occurs in trapezius and scapular area. This typical poster central displacement causes the pain symptoms centrally and bilaterally. Poster lateral movement of disc tissue inserts force on the nerve root, which causes a Segmental pain or root pain and Segmental paraesthesia. Disc displacement may be primary or secondary. Secondary poster lateral displacement is more common type of displacement. Patient previously having pain in different segments like neck, trapezius and scapular region now feels pain in the upper limb area. It occurs due to the lateral shifting of disc tissues.

The goal of treatment in discogenic problems is to stop the conflict between the displaced disc material and affecting sensitive structure. Disc fragment may affect the Dura matter, nerve roots and intervertebral joints. Manipulations and traction brings back the disc material to its place. The choice depends on the displacement. Nuclear displacements are treated by traction while annular ones are by manipulations. Injection usually is done to help pain less spontaneous recovery. If there is too much postero-central displacement that it compresses the spinal cord then surgery usually is done.

Physiotherapy Treatment protocol for cervical discogenic pain include muscle strengthening and to relieve stress on muscles. Cyriax manipulation is a systematic technique of manipulation for the disc prolapse. this study hypothesize that there is a difference between the effects of traditional physical therapy and cyriax manipulation for the discogenic problems. The objecvtive of this study is to find the effects of cyriax manipulation and to compare it with traditional physical therapy treatment in patients with cervical discogenic pain.

Literature review A systematic and evidence based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines. Search term for the initial literature review was discogenic pain, prevalence of neck pain, financial burden of discogenic pain, causes of neck pain, pathophysiology of discogenic pain, treatment options for discogenic pain, manipulation, cyriax manipulation, short term effects of manipulation. The search was limited to papers in English preferably published since 2000 with full text available. Different studies were available regarding cervical manipulation and its effects but limited data was available regarding cyriax manipulation in recent years.

In 2004, previously concluded 33 high quality RCTs in a Cochrane review on mobilization and manipulation of mechanical neck pain. There was strong evidence that mobilization or manipulations when combined with exercises are beneficial for acute or chronic neck pain with or without headache. 3 -11 sessions were compared against placebo.

In literature June 2004, worked to find best evidence in a systematic review on efficacy of spinal manipulation and mobilization for low back pain and neck pain. They showed that there is moderate evidence that spinal manipulative therapy for chronic neck pain is superior when compared to physical therapy and family physician care.

Another randomized controlled trial to correlate the results of manual therapy, physiotherapy, general practitioner care, placebo in treatment of persistent neck and back pain. They took the patients well defined in sub-groups. Physiotherapy included exercises, massage and modalities (heat, ultra-sound, short-wave diathermy). Manual therapy included spine mobilization and manipulation. General practitioner provided analgesics, posture correction, home exercises and bed rest. Placebo consisted of detuned shortwave diathermy and ultra-sound for 10 mines.).Changes in severity of chief complain and functional limitation was main outcome measured by blinded research assistant. Results shows that manual therapy is significantly better than other sub-groups in chronic conditions younger than 40 years of age.

In 2015, in a Cochrane systematic review on mobilization and manipulation on neck pain showed immediate effects of a single manipulation on sub-acute to chronic neck pain. Multiple sessions of cervical manipulations on acute and chronic neck pain produce immediate and long term effects on the pain, function and quality of life.

Howe et al suggested that Manipulation produced a significant immediate improvement in symptoms in those with pain or stiffness in the neck, and pain/paraesthesia in the shoulder, and a nearly significant improvement in those with pain/paraesthesia in the arm/hand.

Study on the non-surgical treatment of cervical radiculopathy suggest manipulation to be very effective and safe in reducing pain, hypo-mobility and disability.

Randomized clinical trial suggest in their current randomized clinical trial that cervical and thoracic thrust manipulation induce similar changes in Pressure Pain Threshold,(PPT) neck pain intensity, and CROM in individuals with bilateral chronic mechanical neck pain.

The combination of manual therapy and manipulation provide better results than manual therapy alone.

Compared intensive training, physiotherapy and manipulation for patients with chronic neck pain after 6 months and 1 year follow up. They found that there was no significant difference between the three treatments. They suggested that as it is not clear whether it is the result of treatment or effect of time. Future studies are necessary to find out the exact treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and confirmed cases of cervical disco genic pain by Weiner's criteria and Cyriax clinical assessment,
* Discogenic cases with pain either in cervico-scapular area, radiating to arm without any neurological symptoms were the main objects of study.

Exclusion Criteria:

* Patients have vertebrobasilar insufficiency (tested by VBI tests),
* Altanto axial instability (tested by sharp purser test),
* Osteoporosis, Rheumatoid arthritis,
* Neuropathies,
* Recent surgeries and neuropathies were excluded from study.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 4th Day
  Changes from base line Northwick disability index was developed first in Northwick Park hospital, England. It was designed to measure the neck pain and disability over time. It consists of 10, five parts sections. At the end, score is calculated by dividing the obtained score by total (50) multiplied by 100. As the driving section was missing in all the female patients, total score was considered as 45 instead of 50.

SECONDARY OUTCOMES:
NPRS | 4th Day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.
ROM Cervical Spine ( Flexion) | 4th Day
  Changes from the Baseline ROM range of Motion of Cervical spine flexion was taken with the Help of Goniometer
ROM Cervical Spine ( extension) | 4th Day
  Changes from the Baseline ROM range of Motion of Cervical spine extension was taken with the Help of Goniometer
ROM Cervical Spine ( Right side flexion) | 4th Day
  Changes from the Baseline ROM range of Motion of Cervical spine right side flexion was taken with the Help of Goniometer
ROM Cervical Spine ( left side Flexion) | 4th Day
  Changes from the Baseline ROM range of Motion of Cervical spine left side flexion was taken with the Help of Goniometer
ROM Cervical Spine ( right rotation) | 4th Day
  Changes from the Baseline ROM range of Motion of Cervical spine right rotation was taken with the Help of Goniometer
ROM Cervical Spine ( left rotation) | 4th Day
  Changes from the Baseline ROM range of Motion of Cervical spine left rotation was taken with the Help of Goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Risbud MV, Shapiro IM. Role of cytokines in intervertebral disc degeneration: pain and disc content. Nat Rev Rheumatol. 2014 Jan;10(1):44-56. doi: 10.1038/nrrheum.2013.160. Epub 2013 Oct 29. PMID 24166242
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Schoenfeld AJ, George AA, Bader JO, Caram PM Jr. Incidence and epidemiology of cervical radiculopathy in the United States military: 2000 to 2009. J Spinal Disord Tech. 2012 Feb;25(1):17-22. doi: 10.1097/BSD.0b013e31820d77ea. PMID 21430568
- [Background] Burkhardt BW, Brielmaier M, Schwerdtfeger K, Oertel JM. Clinical outcome following anterior cervical discectomy and fusion with and without anterior cervical plating for the treatment of cervical disc herniation-a 25-year follow-up study. Neurosurg Rev. 2018 Apr;41(2):473-482. doi: 10.1007/s10143-017-0872-6. Epub 2017 Jun 23. PMID 28646343
- [Background] Phillips FM, Lee JY, Geisler FH, Cappuccino A, Chaput CD, DeVine JG, Reah C, Gilder KM, Howell KM, McAfee PC. A prospective, randomized, controlled clinical investigation comparing PCM cervical disc arthroplasty with anterior cervical discectomy and fusion. 2-year results from the US FDA IDE clinical trial. Spine (Phila Pa 1976). 2013 Jul 1;38(15):E907-18. doi: 10.1097/BRS.0b013e318296232f. PMID 23591659
- [Background] Gross AR, Hoving JL, Haines TA, Goldsmith CH, Kay T, Aker P, Bronfort G; Cervical Overview Group. A Cochrane review of manipulation and mobilization for mechanical neck disorders. Spine (Phila Pa 1976). 2004 Jul 15;29(14):1541-8. doi: 10.1097/01.brs.0000131218.35875.ed. PMID 15247576
- [Background] Quesnele JJ, Triano JJ, Noseworthy MD, Wells GD. Changes in vertebral artery blood flow following various head positions and cervical spine manipulation. J Manipulative Physiol Ther. 2014 Jan;37(1):22-31. doi: 10.1016/j.jmpt.2013.07.008. Epub 2013 Nov 15. PMID 24239451
- [Background] Bronfort G, Haas M, Evans RL, Bouter LM. Efficacy of spinal manipulation and mobilization for low back pain and neck pain: a systematic review and best evidence synthesis. Spine J. 2004 May-Jun;4(3):335-56. doi: 10.1016/j.spinee.2003.06.002. PMID 15125860
- [Background] Koes BW, Bouter LM, van Mameren H, Essers AH, Verstegen GJ, Hofhuizen DM, Houben JP, Knipschild PG. A randomized clinical trial of manual therapy and physiotherapy for persistent back and neck complaints: subgroup analysis and relationship between outcome measures. J Manipulative Physiol Ther. 1993 May;16(4):211-9. PMID 8340715
- [Background] Arnbak B, Jensen TS, Egund N, Zejden A, Horslev-Petersen K, Manniche C, Jurik AG. Prevalence of degenerative and spondyloarthritis-related magnetic resonance imaging findings in the spine and sacroiliac joints in patients with persistent low back pain. Eur Radiol. 2016 Apr;26(4):1191-203. doi: 10.1007/s00330-015-3903-0. Epub 2015 Jul 22. PMID 26194456